CLINICAL TRIAL: NCT03999827
Title: A Pilot Study of the Low Glycaemic Index Diet in Adults With Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STH20468
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Diet Group (Experimental): Adhere to Low Glycaemic Index diet for 52 weeks, beginning immediately after randomisation.
  Interventions: Other: Low Glycaemic Index Diet
- Delayed Diet Group (Active Comparator): Adhere to Low Glycaemic Index diet for 52 weeks, beginning 12 weeks after randomisation.
  Interventions: Other: Low Glycaemic Index Diet

INTERVENTIONS:
Other: Low Glycaemic Index Diet — Adherence to a diet which limits carbohydrate intake to 40-60 g/day, but carbohydrates must have a glycaemic index of less than 50. Fat and protein intake is encouraged, with approximately 60% of calorie intake as fat.
  Other Names: LGI Diet

SUMMARY:
Many persons with epilepsy have seizures which remain uncontrolled by anti-epilepsy medications and are unsuitable for or unwilling to undergo surgical treatments for their epilepsy, or have undergone such treatments and continue to have seizures. Dietary treatments for epilepsy have been shown to be effective in children, and are probably effective in adults, but compliance with the classic ketogenic diet (KD) and to some degree also the modified Atkins diet (MAD) seems difficult for many adults.

The LGI diet may be easier and in children appears to be of comparable efficacy to other dietary treatments (KD and MAD), but has been little studied in adults.

This is a randomised study of immediate versus deferred LGI diet in adults with seizures incompletely controlled by anti-epilepsy medications. 12 weeks of dietary treatment in those randomised to LGI will be followed by the opportunity for the control group to undertake 12 weeks of the LGI diet.

ELIGIBILITY:
Inclusion Criteria:

* adults (>18 years)
* epilepsy refractory to at least two appropriate first line anti-epileptic drugs in adequate dose, unsuitable for or unwilling to undergo surgery for epilepsy.
* At least 1 seizure per week.
* BMI >18

Exclusion Criteria:

* unable to give informed consent
* unable to comply with diet
* surgery for epilepsy or VNS within the last 12 months
* non-epileptic seizures
* pregnant or planning pregnancy
* significant renal impairment
* history of renal stones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
% of patients who adhere to the diet as recorded in food diaries | 52 weeks
  Adherence to the diet will be assessed by self report food diaries which patients will keep. These will be assessed at 12 weeks and 52 weeks after beginning the diet.
Score on diet adherence likert scale questionnaire | 52 weeks
  Adherence to the diet will be assessed by patients scores on a self report likert scale, ranging from 1 (follow the diet all the time) to 5 (follow the diet none of the time), at 12 weeks and 52 weeks after beginning the diet.
Score on diet acceptability likert scale questionnaire | 52 weeks
  Acceptability of the diet will be assessed by patients scores on a self report likert scale, ranging from 1 (the diet is acceptable all of the time) to 5 (the diet is acceptable none of the time), at 12 weeks and 52 weeks after beginning the diet.

SECONDARY OUTCOMES:
Proportion of patients showing a 50% or greater reduction in seizure frequency from baseline | 52 weeks
  Seizure frequency will be assessed through patient completion of seizure diaries throughout the study. This will be assessed at baseline and 12 weeks, 24 weeks and 52 weeks after beginning the diet.
Change from baseline in QOLIE-31 score | 52 weeks
  Epilepsy related quality of life will be measured using the Quality of Life in Epilepsy Inventory-31 (QOLIE-31), a self report questionnaire comprising two factors (emotional and psychological effects, and medical and social effects), eight sub-scales, and 39 items. Items are measured on 4- to 6- point Likert scales, with a maximum total score of 100. Higher scores indicate a better QoL. Change in QOLIE-31 score from baseline to 12 week and 52 weeks after beginning the diet will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Howell, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Royal Hallamshire Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No